CLINICAL TRIAL: NCT01179087
Title: Sleep Disordered Breathing and Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Other Study IDs: B32220109109
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Sleep Disordered Breathing; Lung Transplantation
Keywords: sleep disordered breathing; lung transplantation
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate the prevalence, clinical predictors and consequences (effect on survival, chronic rejection) of sleep disordered breathing in lung transplant recipients.

DETAILED DESCRIPTION:
All patients with end-stage respiratory failure who are referred for lung transplantation and are older than 18 years old are enrolled.

We collect:

* Medical history
* Blood pressure
* Anthropometrics
* Pulmonary function
* Arterial blood gas
* Questionnaire (QOL, ESS)
* Sleep diary
* Polysomnography

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage respiratory failure who are referred for lung transplantation
* Informed consent from patient

Exclusion Criteria:

* Patients who are declined for lung transplantation
* Patients < 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lung transplantation
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disordered breathing | 1 month after lung transplantation
  Polysomnography will be performed at discharge from the hospital (1 month average)
Prevalence of sleep disordered breathing | 1 year after lung transplantation
  Polysomnographic evaluation

SECONDARY OUTCOMES:
Pulmonary function | 1 year after lung transplantation
  Effect of SDB on pulmonary function/BOS
Investigate possible relationship between SDB and patient medical history | 1 year after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bertien MA Buyse, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium